CLINICAL TRIAL: NCT04061356
Title: Assessment of Exhaled Breath Condensate Hydrogen Peroxide (EBC H2O2) as Measured Using a New Device (Inflammacheck™) in Patients With Interstitial Lung Disease, Lung Cancer and Healthy Volunteers. The EXHALE 1B Study
Brief Title: Assessment of Exhaled Breath Condensate Hydrogen Peroxide (EBC H2O2) as Measured Using a New Device (Inflammacheck™) in Patients With Interstitial Lung Disease, Lung Cancer and Healthy Volunteers.
Acronym: EXHALE 1B
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHT/2017/121
Record Dates: First submitted 2019-05-03; First posted 2019-08-19 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Interstitial Lung Disease; Lung Cancer
MeSH Terms: conditions — Lung Diseases, Interstitial; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional study of EBC H2O2 levels, as measured by a novel device, 'Inflammacheck™', and other markers of disease severity in patients with ILD and Lung Cancer.

DETAILED DESCRIPTION:
Inflammation and oxidative stress are processes that occur early in the disease process within both ILD and lung cancer. Current tools for assessing inflammation and oxidative stress, such as fibre-optic bronchoscopy with bronchial wall biopsy and bronchial fluid lavage, are invasive procedures not suitable for regular repeat sampling. Sample analysis requires a series of laboratory measurements and results can take over 24 hours to become available.

In contrast, measurement of Exhaled Breath Condensate Hydrogen Peroxide (EBC H2O2) is performed during normal tidal breathing, and is well tolerated even in patients with severe airways obstruction and those unable to perform a consistent controlled exhalation. It is also not limited to inflammatory cell specific inflammation.

To date, the measurement of EBC H2O2 has been used as a research tool only, due to the complex multiple procedural steps required to deliver a result from the collected exhaled breath. Exhalation Technology Ltd. have now developed a novel, handheld device (Inflammacheck™) which can produce an immediate measurement of EBC H2O2 levels at the patient's side. By detecting EBC H2O2 levels immediately, Inflammacheck™ could tell clinicians and patients the current level of global airway inflammation in a simple, effort independent manner. This could be used by clinicians to diagnose ILD and even Lung Cancer.

The 'Inflammacheck™' device now requires a study in a clinical setting to determine whether it can detect ILD and Lung Cancer. The acceptability and ease of use of the device also needs to be assessed for both patients and clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged ≥18 years.
* A confirmed, clinician made diagnosis of Interstitial Lung Disease (ILD) supported by evidence of ILD on a CT chest scan recorded at any time.
* OR a clinician suspected or confirmed Lung Cancer, with or without asthma and/or COPD
* OR a healthy volunteer with no known history of lung disease (defined as no current clinical diagnosis of, or be receiving treatment for, a lung disease).
* Willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Existing co-morbidities that may prevent them from performing spirometry or other study measurements (at the discretion of the clinical investigator).
* Known other lung, chest wall, neuromuscular, or cardiac disease or abnormality (including end-stage disease or cancer) that would confound symptom scores and spirometry.
* In the opinion of the clinical investigator, participant could be put at risk of harm by having to perform any of the study procedures.
* Unable to comprehend the study and provide informed consent, e.g. insufficient command of English in the absence of someone to adequately interpret.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 75 participants will be recruited, comprised of 50 participants with an established diagnosis that affects their breathing and 25 participants with no history of disease (healthy volunteers).
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-09-14 (Actual); Study Completion 2019-09-14 (Actual)

PRIMARY OUTCOMES:
Level of exhaled breath condensate hydrogen peroxide (EBC H2O2) | 1 day study visit
  Respiratory outcome EBC H2O2 levels as measured by 'Inflammacheck™'

SECONDARY OUTCOMES:
Experience outcome | 1 day study visit
  rating of ease of use of test and participants perception of device as assessed by self completion questionnaire
Disease Stage (lung cancer) | 1 day study visit
  measured by Tumour, Node, Metastasis stage
Disease stage (interstitial lung disease) | 1 day study visit
  measured by the GAP index
safety outcome | 1 day study visit
  incidence of adverse events reported during the study procedures

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No